CLINICAL TRIAL: NCT04441164
Title: VERARE : Effectiveness of Virtual Motor Actions for Improving Walking in Patients With Post-resuscitation Muscle Weakness
Acronym: VERARE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Submitted, denied (too much steps; project to be cut in several projects)
Sponsor: Rennes University Hospital (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC20_8897_VERARE; 2020-A01722-37 (Other: IDRCB)
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Weakness of the Lower Limbs

STUDY DESIGN:
Intervention Model Description: * Step 1: 40 patients (20 in the Virtual Reality group and 20 in the Relaxation group)
  * Step 2: Estimated response rate of approximately 300 caregivers and 50 patients
  * Step 3: 40 patients (20 in the Virtual Reality group and 20 in the Relaxation group)
  * Step 4: 40 patients (20 in the group Performing Virtual Actions and 20 in the group Observing Virtual Actions)
  * Step 5: 40 patients (20 in the group with Haptic stimulation, 20 in the group without Haptic stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Observation of Virtual Actions (steps 1 and 3) (Experimental): If the patient is included in the Virtual Reality group, he/she will be asked to observe Virtual Motor Actions (their own avatar moving in a virtual environment) using a headset once a day for 9 days during 5 minutes, followed by 5 minutes of relaxation performed using soothing music played through headphones.
  Interventions: Other: Observation of Virtual Actions
- Relaxation (Placebo Comparator): If the patient is included in the Relaxation group, he/she will be offered 10 minutes of relaxation performed using soothing music played in headphones once a day for 9 days.
  Interventions: Other: Relaxation
- Patients (Other): It will be offered to patients hospitalized in these 2 services and presenting post-resuscitation ICU-weakness, especially in the aftermath of COVID infection, to complete an acceptability questionnaire (a priori) concerning the use of a Virtual Reality tool intended to improve walking in the ICU. The duration of filling in this questionnaire is estimated at 30 minutes.
  Interventions: Other: Acceptability questionnaire
- Caregivers (Other): It will be offered to caregivers of the ICU of the Rennes University Hospital, to complete an acceptability questionnaire (a priori) concerning the use of a Virtual Reality tool intended to improve walking in the ICU. The duration of filling in this questionnaire is estimated at 30 minutes.
  Interventions: Other: Acceptability questionnaire
- Relaxation (step 3) (Experimental): If the patient is included in the Relaxation group, he/she will be offered 10 minutes of relaxation performed using soothing music played in headphones once a day for 9 days.
  Interventions: Other: Relaxation
- Performing Virtual Actions (Experimental): If the patient is included in the group Performing Virtual Actions, he/she will be asked to perform Virtual Actions of the lower limbs by controlling the legs of his avatar (virtual double) in order to move around in a virtual environment for 10 minutes per day, once a day for 9 days.
  Interventions: Other: Performing Virtual Actions
- Observation of Virtual Actions (Placebo Comparator): If the patient is included in the Observation of Virtual Actions group, he/she will be asked to observe for 10 minutes once a day for 9 days Virtual Motor Actions (avatar moving in a virtual environment) using a Virtual Reality headset.
  Interventions: Other: Observation of Virtual Actions (step 4)
- Haptic stimulation (Experimental): Depending on the superiority or not of the Realization of Virtual Actions or the Observation of Virtual Actions, we will test the most effective condition of step 4 in combination with haptic stimulation (sensory feedback through vibrators positioned in the lower limbs to give a feeling of walking), once a day for 10 minutes for 9 days.
  Interventions: Other: Haptic stimulation
- Without haptic stimulation (Placebo Comparator): Without haptic stimulation Depending on the superiority or not of the Realization of Virtual Actions or the Observation of Virtual Actions, we will test the most effective condition of Step 4 in combination without haptic stimulation (without sensory feedback through vibrators positioned in the lower limbs to give a feeling of walking), once a day for 10 minutes for 9 days.
  Interventions: Other: Without haptic stimulation

INTERVENTIONS:
Other: Observation of Virtual Actions — If the patient is included in the Virtual Reality group, he/she will be asked to observe Virtual Motor Actions (their own avatar moving in a virtual environment) using a headset once a day for 9 days during 5 minutes, followed by 5 minutes of relaxation performed using soothing music played through headphones.
  Arms: Observation of Virtual Actions (steps 1 and 3)
Other: Relaxation — If the patient is included in the Relaxation group, he/she will be offered 10 minutes of relaxation performed using soothing music played in headphones once a day for 9 days.
  Arms: Relaxation; Relaxation (step 3)
Other: Acceptability questionnaire — It will be asked to complete an acceptability questionnaire (a priori) concerning the use of a Virtual Reality tool intended to improve walking in the ICU. The duration of filling in this questionnaire is estimated at 30 minutes.
  Arms: Caregivers; Patients
Other: Observation of Virtual Actions (step 4) — If the patient is included in the Observation of Virtual Actions group, he/she will be asked to observe for 10 minutes once a day for 9 days Virtual Motor Actions (avatar moving in a virtual environment) using a Virtual Reality headset.
  Arms: Observation of Virtual Actions
Other: Performing Virtual Actions — If the patient is included in the group Performing Virtual Actions, he/she will be asked to perform Virtual Actions of the lower limbs by controlling the legs of his avatar (virtual double) in order to move around in a virtual environment for 10 minutes per day, once a day for 9 days.
  Arms: Performing Virtual Actions
Other: Haptic stimulation — According to the superiority or not of the Realization of Virtual Actions or the Observation of Virtual Actions, we will test the most effective condition of step 4 in combination with haptic stimulation (sensory feedback through vibrators positioned in the lower limbs to give a feeling of walking), once a day for 10 minutes for 9 days.
  Arms: Haptic stimulation
Other: Without haptic stimulation — Without haptic stimulation Depending on the superiority or not of the Realization of Virtual Actions or the Observation of Virtual Actions, we will test the most effective condition of Step 4 in combination without haptic stimulation (without sensory feedback through vibrators positioned in the lower limbs to give a feeling of walking), once a day for 10 minutes for 9 days.
  Arms: Without haptic stimulation

SUMMARY:
After a hospitalization in Intensive Care Unit (ICU), approximately 50% of patients usually have a ICU-Weakness, i.e. nerves and muscles injury secondary to immobilization and to treatments which had to be used. This disease is expected to be similar or even higher in patients suffering from COVID-19 and hospitalized in ICU due to the average length of hospitalization of several weeks in this population. This condition will delay the return-to-walk of these patients, their discharge from hospitalization and may deteriorate their autonomy in daily life activities.

Virtual Reality (VR) environments are already used and have proven their worth for the assessment and rehabilitation of patients with neurological diseases. It therefore seems appropriate to offer the use of virtual environments for this type of population. VR represents a unique opportunity for the rehabilitation care of these patients, and in particular those who have been reached by COVID-19, due to the possible mismatch between the amount of motor rehabilitation to be provided and the fatigability and breathlessness at the slightest effort which seem particularly intense in this population.

The main objective of our project is to improve and to accelerate gait recovery in patients hospitalized in Physical and Rehabilitation Medicine after discharge from Resuscitation or Continuous Care Unit and in patients hospitalized in ICU and presenting ICU-weakness secondary to resuscitation, notably due to COVID-19 infection, thanks to the use of Virtual Reality tools. The VR tool will consist of virtual environments presented using a Virtual Reality headset where an avatar (double) of the patient hospitalized in Physical and Rehabilitation Medicine or in ICU will be represented, who will perform different motor tasks involving their lower limbs (ex: walking, or kicking a ball) in several different virtual environments (settings). The patient will be asked to observe actions, then to imagine carrying out their actions which will be performed by the avatar in the virtual environment, then they will be able to control the actions of the avatar using their legs thanks to sensors, then feel walking sensations through the use of haptic devices.

DETAILED DESCRIPTION:
Step 1: The objective is to evaluate the effectiveness of the Observation of Virtual Actions on gait recovery in patients hospitalized in Physical and Rehabilitation Medicine (MPR) and presenting ICU-weakness, in particular following a COVID-19 infection. If the patient is included in the Virtual Reality group, they will be asked to observe once a day for 9 days for 5 minutes Virtual Motor Actions (avatar moving in a virtual environment) using a headset. Virtual Reality, followed by 5 minutes of relaxation performed using soothing music played through headphones. If the patient is included in the Relaxation group, they will be offered 10 minutes of relaxation performed using soothing music played in headphones once a day for 9 days. We will assess gait, motive power, balance, confidence in the future and patient autonomy before the start of the first session, the day after the last session and one month after inclusion. At the end of each session, we will ask the patient questions about fatigue (VAS) and the occurrence of side effects (open question) after wearing the Virtual Reality headset or headset. At the end of the 9 sessions, we will ask to patients in the Virtual Reality group to complete a questionnaire concerning the acceptance of the proposed device. We want to include 20 patients in the Virtual Reality group and 20 patients in the Relaxation group.

Step 2: The objective is to assess the acceptability (a priori) of the Virtual Reality tool created in ICU by the nursing staff and by the patients who are hospitalized there. It will be offered to caregivers of the ICU of the Rennes University Hospital and to patients hospitalized in these 2 services and presenting ICU- weakness, especially in the aftermath of COVID infection. We will be asked to complete an acceptability questionnaire (a priori) concerning the use of a Virtual Reality tool intended to improve walking in the ICU. The duration of filling in this questionnaire is estimated at 30 minutes. Caregivers will be invited to participate in an information meeting (4 will be carried out) at least 1 week before their possible participation (which they will be informed by internal mail, and which will be led by investigators). We believe that approximately 300 caregivers and 50 patients will participate in this acceptability survey.

Step 3: The objective is to evaluate the effectiveness of the Observation of Virtual Actions on gait recovery in patients hospitalized in ICU and with ICU-weakness. If the acceptability questionnaire is in favor of a good future acceptance of the tool designed and after possible adaptations of the Virtual Reality device based on the responses of caregivers and patients to the acceptability questionnaire proposed during the step 2, we will suggest to patients hospitalized in ICU with ICU-weakness to carry out a protocol similar to that carried out with Physical and Rehabilitation Medicine patients in step 1. If the patient is included in the Virtual Reality group, they will be asked to observe once a day for 9 days for 5 minutes Virtual Motor Actions (avatar moving in a virtual environment) using a Virtual Reality headset, followed by 5 minutes of relaxation performed using soothing music played through headphones. If the patient is included in the Relaxation group, they will be offered 10 minutes of relaxation performed using soothing music played in headphones once a day for 9 days. We will assess gait, motive power, balance, confidence in the future and patient autonomy before the start of the first session, the day after the last session and 1 month after inclusion. At the end of each session, we will ask the patient questions about fatigue (VAS) and the occurrence of side effects (open question) after wearing the Virtual Reality headset. At the end of the 9 sessions, we will suggest to patients in the Virtual Reality group that they complete a questionnaire concerning the acceptance of the proposed device. We want to include 20 patients in the Virtual Reality group and 20 patients in the Relaxation group.

Step 4: The objective is to assess the effectiveness of the realization of virtual actions compared to the observation of virtual actions on gait recovery in patients hospitalized in ICU or in Physical and Rehabilitation Medicine and presenting ICU-weakness. If the patient is included in the group Performing Virtual Actions, they will be asked to perform Virtual Actions of the lower limbs by controlling the legs of his avatar (virtual double) in order to move around in a virtual environment for 10 minutes per day, once a day for 9 days. If the patient is included in the Observation of Virtual Actions group, they will be asked to observe for 10 minutes once a day for 9 days Virtual Motor Actions (avatar moving in a virtual environment) using a Virtual Reality headset. We will assess gait, motive power, balance, confidence in the future and patient autonomy before the start of the first session, the day after the last session and 1 month after inclusion. At the end of each session, we will ask the patient questions about fatigue (VAS) and the occurrence of side effects (open question) after wearing the Virtual Reality headset. At the end of the 9 sessions, we will offer patients to fill out a questionnaire concerning the acceptance of the proposed device. We want to include 20 patients in the Virtual Actions group and 20 patients in the Virtual Actions Observation group.

Step 5: The objective is to evaluate the effectiveness of adding a sensation of walking using haptic stimuli during the Observation or Realization of Virtual Actions on the recovery of walking in patients hospitalized in ICU or in Physical and Rehabilitation Medicine and with ICU-weakness. Depending on the superiority or not of the Realization of Virtual Actions or the Observation of Virtual Actions, we will test the most effective condition of step 4 in combination with: either haptic stimulation (sensory feedback through vibrators positioned on the lower limbs to give a feeling of walking), either without haptic stimulation, once a day for 10 minutes for 9 days. We will assess gait, motive power, balance, confidence in the future and patient autonomy before the start of the first session, the day after the last session and 1 month after inclusion. At the end of each session, we will ask the patient questions about fatigue (VAS) and the occurrence of side effects (open question) in the aftermath of wearing a Virtual Reality headset. At the end of the 9 sessions, we will offer patients to fill out a questionnaire concerning the acceptance of the proposed device. We want to include 20 patients in the group with haptic stimulation and 20 patients in the group without haptic stimulation.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Step 1: Patient hospitalized in the Physical Medicine and Rehabilitation department of the Rennes University Hospital following a stay in intensive care or in a Continuing Care Unit, in particular following a COVID-19 infection, and with muscle weakness of the lower limbs with an MRC motor testing on the main muscle segments giving a score less than or equal to 48/60 (diagnostic criterion of ICU Weakness)
* Steps 2 and 3: Patient hospitalized in one of the ICU of the Rennes University Hospital and presenting post-resuscitation muscle weakness in the lower limbs with MRC motor testing on the main muscle segments giving a score less than or equal to 48/60 (diagnostic criterion of ICU Weakness)
* Steps 4 and 5: Patient hospitalized in one of the ICU or in the Physical Medicine and Rehabilitation service of the Rennes University Hospital and presenting post-resuscitation muscle weakness in the lower limbs with an MRC motor testing on the main muscle segments giving a score less than or equal to 48/60 (diagnostic criterion of ICU-Weakness)

For nursing staff:

Step 2: Person with one of the following professions: nursing assistant, nurse, doctor, physiotherapist, and practicing for more than a month in one of the ICU of the Rennes University Hospital .

For everyone :

* Person of full age;
* Affiliation to a social security insurance;
* Free, informed and written consent signed.

Exclusion Criteria:

For patients:

* History of central neurological event with clinical repercussions;
* Gait disturbances preexisting in ICU hospitalization and limiting the gait perimeter (declaration by the patient) or requiring the use of technical assistance;
* Uncontrolled epilepsy (last crisis occurring less than 6 months old);
* Persons of full age subject to legal protection (safeguard of justice, curators, guardians), persons deprived of their liberty;
* Pregnant or lactating woman.

For caregivers:

* Non-French fluent people;
* Adults over the age of legal protection (safeguard of justice, curators, guardians), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
6-minute test | Day 10
  Number of meters taken during the 6-minute test the day after the last session.

SECONDARY OUTCOMES:
Time for 10-meter test | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Gait assessment before the start of the first session, the day after the last session and 1 month from inclusion: 10-meter test (time in seconds)
6-minute walk test | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Gait assessment before the start of the first session, the day after the last session and 1 month from inclusion: 6-minute walk test (need for breaks, scale de Borg, existence of desaturation)
Recovery time | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Gait assessment before the start of the first session, the day after the last session and 1 month from inclusion: recovery time for walking over 10 meters without human or technical assistance
Normal or deficient posture balance in sitting and standing | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Assessment of balance before the start of the first session, the day after the last session and 1 month from inclusion: normal or deficient posture balance in sitting and standing
Berg Balance Scale | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Assessment of balance before the start of the first session, the day after the last session and 1 month from inclusion: Berg Balance Scale. Berg's balance scale includes 14 tests that assess static balance and dynamic balance. Each test is rated from 0 (needs help) to 4 (can do on him/her own). Total score is on 56 points.
Timed Up and Go test | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Assessment of balance before the start of the first session, the day after the last session and 1 month from inclusion: Timed Up and Go test (time in seconds)
Duration for the test of the 10 chair lifts | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Assessment of balance before the start of the first session, the day after the last session and 1 month from inclusion: test of the 10 chair lifts (duration in seconds, existence of a desaturation, Borg scale)
MRC scale | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Strength assessment before the start of the first session, the day after the last session and within 1 month of inclusion: MRC testing of the lower limbs.
  The Medical Research Council's scale (MRC scale) is an assessment of muscle power, rated form 0 (no contraction) to 5 (normal power).
Functional Independence Measure | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Assessment of autonomy before the start of the first session, the day after the last session and within 1 month of inclusion: Functional Independence Measure.
  The Functional Independence Measure (FIM) is an 18-item instrument measuring a person's level of disability in terms of burden of care. Each item is rated from 1 (requiring total assistance) to 7 (completely independent). Three independent FIM scores can be generated by summing item scores: a total score (FIM total: 18 items), a motor score (FIM motor: eating, grooming, bathing, dressing - upper body, dressing - lower body, toileting, bladder management, bowel management, and transfers bed/chair/wheelchair, toilet, tub/shower, walk, stairs), and a cognitive score (FIM cognitive: auditory comprehension, verbal expression, social interaction, problem solving, and memory). Multiple studies support the reliability and validity of FIM scales in the older population.
Acceptability | Day 1 (step 2)
  Acceptability (a priori, patients and caregivers for stage 2) questionnaires
Acceptance | Day 1 (step 2)
  Acceptance (patients for stages 1, 3, 4 and 5) questionnaires
Fatigue | End of each session, at days 1 to 9
  Fatigue assessment (visual analog scale) (steps 1, 3, 4, 5)
Undesirable effects | End of each session, at days 1 to 9
  Collections of possible undesirable effects by open question at the end of each session with the Virtual Reality tool (steps 1, 3, 4, 5)
Confidence in the future | Before the start of the first session (day 1), the day after the last session (day 9) and 1 month after inclusion
  Assessment of confidence in the future using a questionnaire (steps 1, 3, 4, 5) before the start of the first session, the day after the last session and 1 month from inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No